CLINICAL TRIAL: NCT01617824
Title: Rapid Effects of the DPP-4 Inhibitor Linagliptin on Monocyte Polarization and Endothelial Progenitor Cells in Type 2 Diabetic Patients With and Without Chronic Renal Failure. A Randomized Cross-over Trial Versus Placebo
Brief Title: Rapid Effects Linagliptin on Monocyte Polarization and Endothelial Progenitor Cells in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2588P
Record Dates: First submitted 2012-06-03; First posted 2012-06-12 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes; Chronic Renal Failure
Keywords: Diabetes; Kidney; Inflammation; Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Diabetes Mellitus; Inflammation | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin (Experimental): Linagliptin 5 mg tablets daily for 4 days
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Placebo tablets 1 daily for 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin — Linagliptin 5 mg tablets for 4 days
  Other Names: Trajenta 5 mg
  Arms: Linagliptin
Drug: Placebo — Placebo tablets for 4 days
  Arms: Placebo

SUMMARY:
Diabetes mellitus is characterized by chronic low grade inflammation, which is worsened by the co-existence of renal failure.

One key aspect of chronic inflammatory diseases is the alteration in the polarization profile of circulating monocyte-macrophage cells.

Namely, monocytes-macrophages can exist in a pro-inflammatory (M1) polarized form or an anti-inflammatory (M2) polarized state. Alterations in the M1/M2 balance is thought to contribute to inflammation within atherosclerotic lesions and visceral adipose tissue which, in turn, can worsen cardiovascular disease and metabolic features in type 2 diabetic patients.

M1 and M2 are regulated by a complex interplay of soluble signaling molecules, many of which are substrate of the enzyme DPP-4 (dipeptidyl peptidase-4). Therefore, inhibition of DPP-4 can affect the M1/M2 polarization balance.

In this clinical trial, the investigators will test whether the DPP-4 inhibitor Linagliptin, compared to placebo, modifies the M1/M2 balance in type 2 diabetic patients with and without chronic renal failure.

In addition, we will test whether DPP-4 inhibition with Linagliptin acutely affects endothelial progenitor cells (EPCs), which are vasculoprotective cells implicated in the pathobiology of diabetic complications.

DETAILED DESCRIPTION:
Type 2 diabetes is associated with chronic sterile low-grade inflammation, usually caused by hyperglycemia and associated biochemical abnormalities, as well as by overweight/obesity. The co-existence of chronic renal failure further exacerbates inflammation in diabetic patients, and this contributes to the exceedingly high morbidity and mortality of this category of patients. One key element of this type of inflammation is the pro- versus anti-inflammatory polarization of circulating monocytes and tissue macrophages. Diabetes indeed causes an imbalance of this polarization, in favour of the pro-inflammatory (M1) monocytes at the expenses of anti-inflammatory (M2) monocytes. Cells belonging to the monocyte/macrophage lineage are of great importance in diabetes pathophysiology, as they are involved in atherosclerosis and adipose tissue biology, both of which determine diabetes outcomes. It is recognized that M1/M2 polarization relies on the expression of chemokines/cytokines and their respective receptors. Interestingly, among non-incretin substrates of DPP-4 are several chemokines (e.g. MCP-1 and -2, RANTES and SDF-1a), which may regulate M1/M2 polarization. Linagliptin (terminal half-life >100 hours, and effective half-life for accumulation approximately 12 hours) can be safely used in type 2 diabetic patients with renal impairment without dose adjusting, because the drug is excreted >90% with feces and has a minor renal excretion. The possibility to modulate the M1/M2 inflammatory pathway with the DPP-4 inhibitor linagliptin entails a hitherto unappreciated opportunity for protecting diabetic patients with renal disease from the detrimental consequences of chronic inflammation on vascular and adipose tissue biology. We have set up a protocol to assess M1/M2 polarization of circulating monocyte/macrophage cells by flow cytometry. Our preliminary data indicate that diabetes is associated with an imbalance in M1/M2 polarization versus non diabetic controls, in favour of M1 cells in diabetic patients. Hyperglycemia per se may affect M1/M2 polarization and it is expected that any effect of linagliptin on monocytes can be detected as soon as DPP-4 inhibition reaches steady-state. Therefore, in order to provide a proof-of-concept for the effect of linagliptin on M1/M2 polarization and to avoid the confounding of improved glucose control, the time point of the study will be very short (4 days). Our preliminary data in cell cultures indicate that a few days of treatment with a stimulus is sufficient to modulate monocyte/macrophage polarization. This will provide valuable information on the direct effects of the drug on this inflammatory pathway.

Endothelial progenitor cells (EPCs) are vasculoprotective cells released from the bone marrow (BM) in response to ischemia, hypoxia and tissue injury. Once in the bloodstream, EPCs home to damaged tissues and help restoring a healthy and functional vasculature, by means of endothelial repair and angiogenesis. In steady-state conditions, CD34+KDR+ EPCs circulate in peripheral blood (PB) at very low levels and their release from the BM is coordinated by the sympathetic nervous system. It has been demonstrated that levels of EPC and generic CD34+ PC are predictors of future cardiovascular events, cardiovascular death and all-cause mortality. We have previously shown that Sitagliptin raised EPCs levels in 4 weeks. Herein, we aim to confirm those findings using Linagliptin, with a shorter time point.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* eGFR > 60 mL/min/1.73 mq (for the patients without renal failure)
* eGFR 10-60 mL/min/1.73 mq (for the patients with renal failure)

Exclusion Criteria:

* Type 1 diabetes
* Hypersensitivity to Linagliptin or excipients
* Intolerance to other DPP-4 inhibitors
* Terminal renal failure (eGFR < 10 mL/min/1.73 mq)
* Use of GLP-1 analogs or other DPP-4 inhibitors
* Recent (within 1 month) trauma or surgery or acute diseases
* Any acute or chronic inflammatory condition
* Immunosuppression or organ transplantation
* Pregnancy or lactation
* Inability to provide informed consent.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
M1/M2 polarization balance | day 5
  Evaluate whether 4-days Linagliptin treatment, compared to placebo, significantly reduces the M1/M2 ratio in type 2 diabetic patients. In this cross-over design trial, Linagliptin and placebo will be administered once daily for 4 consecutive days to 30 type 2 diabetic patients with or without renal failure with a 2 week washout period in between.

SECONDARY OUTCOMES:
Cytokine and chemokine concentrations | day 5
  Evaluate whether 4-days Linagliptin treatment, compared to placebo, significantly modifies the concentrations of selected cytokines and chemokines (MCP-1, RANTES, SDF-1a, IL-1, IL-6, TNF-a, IL-10, TGF-beta, CCL22, fraktalkine) in type 2 diabetic patients. In this cross-over design trial, Linagliptin and placebo will be administered once daily for 4 consecutive days to 30 type 2 diabetic patients with and without renal failure with a 2 week washout period in between. As the number of measures is high and there is no adjustment for multiple testing, this outcome is to be considered exploratory.
Endothelial progenitor cell levels | day 5
  Evaluate whether 4-days Linagliptin treatment, compared to placebo, significantly modifies the levels of CD34+KDR+ EPCs (outcome added in course)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Avogaro, M.D. Ph.D., Study Chair — University of Padova; Gian Paolo Fadini, M.D., Principal Investigator — University of Padova
Locations (1):
- University Hospital Diabetes Outpatient Clinic, Padua, Italy

REFERENCES:
- [Derived] Fadini GP, Bonora BM, Albiero M, Zaninotto M, Plebani M, Avogaro A. DPP-4 inhibition has no acute effect on BNP and its N-terminal pro-hormone measured by commercial immune-assays. A randomized cross-over trial in patients with type 2 diabetes. Cardiovasc Diabetol. 2017 Feb 10;16(1):22. doi: 10.1186/s12933-017-0507-9. PMID 28183314
- [Derived] Fadini GP, Bonora BM, Cappellari R, Menegazzo L, Vedovato M, Iori E, Marescotti MC, Albiero M, Avogaro A. Acute Effects of Linagliptin on Progenitor Cells, Monocyte Phenotypes, and Soluble Mediators in Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Feb;101(2):748-56. doi: 10.1210/jc.2015-3716. Epub 2015 Dec 22. PMID 26695864